CLINICAL TRIAL: NCT06107673
Title: A Phase II Randomized, Non-inferiority Study Comparing the Efficacy and Safety of Dalpiciclib Combined With AI With Neoadjuvant Chemotherapy in ER+ HER2- Postmenopausal Breast Cancer Patients
Brief Title: Dalpiciclib Plus AI (Neoadjuvant Endocrine Therapy) Compared With Neoadjuvant Chemotherapy in Early Breast Cancer （EBC）
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MA-BC-II-055
Record Dates: First submitted 2023-08-20; First posted 2023-10-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: HER2- ER+; Neoadjuvant therapy; Dalpiciclib
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; Aromatase Inhibitors; Docetaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant endocrine group (Experimental): Dalpiciclib: Take 125 mg once daily for 3 weeks, then stop for 1 week. Each cycle is completed in 4 weeks.
  AI: Take according to the instructions provided.
  Interventions: Drug: Dalpiciclib; Drug: Aromatase inhibitor
- neoadjuvant chemotherapy group (Active Comparator): Docetaxel for injection: Administered as a 75 mg/m2 intravenous infusion Epirubicin hydrochloride for injection: Administered as a 75 mg/m2 intravenous infusion.
  Cyclophosphamide for injection: Administered as a 500 mg/m2 intravenous infusion.
  Interventions: Drug: Docetaxel injection; Drug: Epirubicin Hydrochloride Injection; Drug: Cyclophosphamide injection

INTERVENTIONS:
Drug: Dalpiciclib — Dalpiciclib: Take 125 mg once daily for 3 weeks, then stop for 1 week. Each cycle is completed in 4 weeks. It is recommended to take the medication approximately at the same time each day, with warm water, preferably on an empty stomach. Fasting for at least 1 hour before and after medication is advised.
  Other Names: SHR6390
  Arms: neoadjuvant endocrine group
Drug: Aromatase inhibitor — AI: Take according to the instructions provided.
  Other Names: AI
  Arms: neoadjuvant endocrine group
Drug: Docetaxel injection — Administered as a 75 mg/m2 intravenous infusion over approximately 30 minutes. It is given every three weeks and dose reduction or treatment delay is allowed, up to a maximum delay of 3 weeks from the previous dose calculation. Treatment will be terminated if the delay exceeds this limit.
  Arms: neoadjuvant chemotherapy group
Drug: Epirubicin Hydrochloride Injection — Administered as a 75 mg/m2 intravenous infusion. It is given every three weeks and dose reduction or treatment delay is allowed, up to a maximum delay of 3 weeks from the previous dose calculation. Treatment will be terminated if the delay exceeds this limit.
  Arms: neoadjuvant chemotherapy group
Drug: Cyclophosphamide injection — Administered as a 500 mg/m2 intravenous infusion. It is given every three weeks and dose reduction or treatment delay is allowed, up to a maximum delay of 3 weeks from the previous dose calculation. Treatment will be terminated if the delay exceeds this limit.
  Arms: neoadjuvant chemotherapy group

SUMMARY:
This study is a multi-center, randomized, prospective phase II clinical trial aimed at exploring and evaluating the efficacy of dalpiciclib combined with AI in neoadjuvant treatment for ER strong positive（ER≥50%），HER2-negative, Ki-67≤20%,T1-3N1M0 postmenopausal breast cancer. The primary objectives are to demonstrate non-inferiority in efficacy compared to chemotherapy and to assess its superior safety profile.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, prospective non-inferiority exploratory phase II clinical trial. Eligible subjects were randomly assigned in a 1:1 ratio to either the dalpiciclib combined with AI group （neoadjuvant endocrine group） or the AC-T group （chemotherapy group） after screening. The administration of the investigational drugs started within 48 hours after randomization. Subjects will receive either 24 weeks of dalpiciclib combined with AI or AC-T treatment until disease progression, intolerable adverse events, withdrawal of informed consent, or discontinuation by the investigator's judgment.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form to participate in the clinical research.
2. Confirmed postmenopausal females diagnosed with invasive breast cancer.
3. Clinical stage T1-3N1M0.
4. Pathological examination confirmed: Strong positive for ER, negative for HER2. HER2 negative: Immunohistochemistry (IHC) suggests HER2 (-, +) or (++) but in situ hybridization (ISH) indicates negative. Strong positive for ER: ER immunohistochemistry test shows 50% or more tumor cells positive.
5. No prior breast cancer-related treatment.
6. No concurrent cardiac diseases, baseline left ventricular ejection fraction (LVEF) ≥ 50%, no significant cardiac diseases (≤ NYHA class I).
7. ECOG score of 0-1, meeting the indications and basic requirements for chemotherapy without major organ dysfunction.
8. Within 1 week prior to enrollment, routine blood tests are essentially normal: Absolute neutrophil count (NEUT#) ≥ 1.5×10^9 /L; White blood cell count (WBC) ≥ 3.0×10^9 /L; Platelets ≥ 90×10^9 /L; Hemoglobin ≥ 90 g/L.
9. Within 1 week prior to enrollment, liver and kidney function tests are essentially normal: Total bilirubin (TBIL) ≤ 1.5× upper limit of normal (ULN); Alanine aminotransferase and aspartate aminotransferase (ALT/AST) ≤ 2× ULN; Serum creatinine ≤ 1.5× ULN or creatinine clearance rate (Ccr) ≥ 60 ml/min.
10. For women of childbearing age, negative serum or urine pregnancy test results before participation; premenopausal women during the study period should use medically acceptable methods of contraception.
11. Exhibits good compliance.

Exclusion Criteria:

1. Pregnant or lactating women, and women of childbearing age who have a positive pregnancy test at baseline and do not agree to use effective contraception during the study.
2. Patients with a known history of severe allergic reactions to any investigational drug components (NCI-CTCAE Grade > 3) or with any clearly documented drug allergy.
3. Patients with bilateral breast cancer or inflammatory breast cancer.
4. Patients with metastatic (stage IV) breast cancer at initial diagnosis.
5. Patients with a history of congestive heart failure, unstable angina, arrhythmias, or myocardial infarction.
6. Current diagnosis of acute lung conditions, interstitial lung disease, pulmonary fibrosis, acute pulmonary disease, etc.
7. Current diagnosis of severe liver-related diseases such as acute hepatitis, fulminant hepatitis, coagulation factor synthesis disorders. If HBV surface antigen or HBV core antibody are positive, the peripheral blood HBV DNA titer should be < 1×10^3 IU/ml for eligibility.
8. Any other serious medical condition or comorbidity that may interfere with participation in the study or may significantly affect the safety of the subject (e.g., active or uncontrolled infections, active or requiring antiviral therapy for liver and bile diseases).
9. Other invasive malignancies (including second primary breast cancer) that may interfere with the evaluation of study endpoints and compliance with the protocol.
10. Patients with a history of prior treatment with chemotherapy, endocrine therapy, or anti-HER2 biologic therapy for breast cancer (excluding diagnostic biopsy for primary breast cancer).
11. Patients who have undergone major surgery within 4 weeks prior or have significant unresolved medical conditions.
12. Patients with non-measurable tumors during treatment.
13. Any other condition that the investigator deems unsuitable for the participation of the subject in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Complete Radiologic Response or Partial Radiological Response: Radiological Response | 6 months
  Radiological response is the percentage of participants with CR or, PR according to RECIST v.1.1. A responder is defined as any participant who exhibits a CR or PR. CR is the disappearance of all target lesions. PR is a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. PD is 20% increase in the sum of diameters of target lesions taking as reference the smallest sum and the appearance of 1 or more new lesions.

SECONDARY OUTCOMES:
Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | 6 months
  EORTC QLQ-C30 v3.0 was a self-administered questionnaire with multidimensional scales that measures 5 functional domains (physical, role, emotional, cognitive, or social functioning), global health status and symptom scales of fatigue, pain, nausea/vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, or financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, higher scores represent a better level of functioning. For symptoms scales, higher scores represented a greater degree of symptoms.
Evaluation of the number of patients with a Residual Cancer Burden (RCB) 0-I index | 6 months
  Residual cancer burden (RCB) is estimated from routine pathologic sections of the primary breast tumor site and the regional lymph nodes after the completion of neoadjuvant therapy. 6 variables are included in a calculation formula.
Evaluation of the number of patients with PEPI 0 | 6 months
  PEPI stands for Preoperative Endocrine Prognostic Index. It is a scoring system used in breast cancer research to assess the response to neoadjuvant endocrine therapy. PEPI evaluates various factors, including tumor size, lymph node involvement, Ki-67 proliferation index, and estrogen receptor status, to predict the risk of recurrence and overall prognosis in patients with hormone receptor-positive breast cancer. The PEPI score helps in determining the effectiveness of neoadjuvant endocrine therapy and guiding treatment decisions.
Percentage of Participants With Pathologic Complete Response (pCR) | 6 months
  pCR is defined as absence of invasive cancer in the breast and sampled regional lymph nodes.
Calculation of the rates of breast conservation therapy in the two arms with regard to the initially planned surgery. | 6 months
Percent Change From Baseline to 2 Weeks in Ki67 Expression | 2 Weeks
  Tumor tissue collected through a core biopsy at baseline and at the end of cycle 1 was used to determine Ki67 expression. Ki67 expression is defined as the percent of cells staining positive by validated central assay.
Determination of the number and type of Adverse Events as a Measure of Safety and Tolerability | 6 months
  The toxicity will be evaluated according to the scale CTC-AE version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No